CLINICAL TRIAL: NCT00004695
Title: Randomized Study of Polyethylene-Glycol-Conjugated Interleukin 2 in Patients With Common Variable Immunodeficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: 199/13358; MTS-93-726-ME; MTS-FDR001162
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 1999-05

CONDITIONS: Common Variable Immunodeficiency
Keywords: common variable immunodeficiency; immunologic disorders and infectious disorders; primary immunodeficiency disease; rare disease
MeSH Terms: conditions — Common Variable Immunodeficiency; Immune System Diseases; Communicable Diseases; Primary Immunodeficiency Diseases; Rare Diseases | interventions — interleukin-2, polyethylene glycol-modified

INTERVENTIONS:
Drug: PEG-interleukin-2

SUMMARY:
OBJECTIVES: I. Determine whether polyethylene-glycol-conjugated interleukin 2 (PEG-IL-2) can reduce the number of infections in patients with common variable immunodeficiency.

II. Determine whether this therapy can improve lung functions in these patients with pulmonary impairment.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, open-label study. Patients are randomized to receive polyethylene-glycol-conjugated interleukin 2 (PEG-IL-2) or placebo.

Patients receive PEG-IL-2 or placebo by subcutaneous injection weekly for 18 months. Patients maintain a daily diary for 24 months.

Patients are followed every 4 months for 2 years.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Documented common variable immunodeficiency defined as a reduction of serum IgG by at least 2 standard deviations

In vitro lymphocyte proliferative response to PEG-IL-2 of at least 10 times more than unstimulated cultures

--Prior/Concurrent Therapy--

No biologic response modifier therapy (i.e., interferon, cyclosporin A) except prednisone (maximum 10 mg/day)

Concurrent treatment with same dosage intravenous gamma-globulin for at least 6 months is required

--Patient Characteristics--

Life expectancy: At least 24 months

Other: Not pregnant or nursing HIV negative

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48
Dates: Start 1997-09; Study Completion 2000-03

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Cunningham-Rundles, Study Chair — Icahn School of Medicine at Mount Sinai